CLINICAL TRIAL: NCT03422367
Title: Mechanisms of Change With Early Intervention in Tuberous Sclerosis
Brief Title: JASPER Early Intervention for Tuberous Sclerosis
Acronym: JETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Boston Children's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Shafali Jeste, MD, Director of Developmental Neurophysiology Lab, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #17-000262; 1R01HD090138-01A1 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Tuberous Sclerosis
Keywords: autism; epilepsy; asd; TSC; UCLA; Los Angeles; JASPER; intervention; Boston; BCH; MGH
MeSH Terms: conditions — Tuberous Sclerosis; Autistic Disorder; Epilepsy; Child Development Disorders, Pervasive | interventions — Activator Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): The Treatment Group begins the JASPER intervention immediately upon enrollment in the study.
  Interventions: Behavioral: JASPER
- Delayed Treatment Group (Active Comparator): The Delayed treatment group receives the same JASPER intervention as the Treatment Group, but after 6 months of receiving services in the community as usual.
  Interventions: Behavioral: JASPER
- Control (No Intervention): Participants who are unable to complete JASPER due to age or time/distance commitment can enroll for single-time point participation

INTERVENTIONS:
Behavioral: JASPER — JASPER (Joint Attention, Symbolic Play, Engagement, and Regulation) is a treatment approach based on a combination of developmental and behavioral principles developed by Dr. Connie Kasari and Dr. Amanda Gulsrud at UCLA. It targets the foundations of social communication (joint attention, imitation, play) and uses naturalistic strategies to increase the rate and complexity of social communication.
  Other Names: Joint Attention; Symbolic Play and Engagement Regulation
  Arms: Delayed Treatment Group; Treatment Group

SUMMARY:
The investigators are running an intervention study for young children with Tuberous Sclerosis Complex (TSC). The study will include free play-based behavioral intervention administered remotely that may improve social and communication skills in children with TSC. Eligible families will have a child in the age range of 12-36 months, with a diagnosis of TSC. Children with TSC below 12 months may be eligible for an early markers study prior to enrollment in the intervention trial.

The intervention will focus on teaching caregivers skills to improve the social and communication outcomes of their children. The content of the intervention will be individually tailored to the child's developmental level. The intervention involves 4 on-site assessment visits, and 12 weekly intervention sessions, administered in-person and remotely. The intervention focuses on improving social-communication and play skills.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is a genetic disorder caused by mutations in either the TSC1 or TSC2 genes. The genetic variation results in the growth of non-malignant tumors throughout the body. Neurodevelopmental disorders, including global developmental delay, intellectual disability, and autism spectrum disorder (ASD) are very common in children with TSC, although developmental outcomes can vary widely. Study investigators, over the past several years, has been studying infants and young children with TSC, and investigators have found that developmental delays can be identified in the first year of life, and that these delays and differences can predict a diagnosis of ASD. Currently, there is no specific treatment for the neurodevelopmental disorders associated with TSC. Based on this information, researchers now want to know if early intervention can help to improve development and prevent ASD in children with TSC.

Investigators are studying the effects of early behavioral intervention on developmental outcomes in infants and toddlers with TSC. The study focuses on social-communication skills, as these are tightly linked to the development of ASD. The overarching goal of this research is to improve outcomes in infants with TSC by conducting rigorous, innovative research in treatment, using both brain and behavioral measures to study the effects of treatment.

Participation requires four on-site assessment visits at UCLA or Boston Children's Hospital, and 12 weekly behavioral intervention sessions, administered in-person and remotely. Because this behavioral intervention is parent-mediated, a parent must be available to attend these sessions. Behavioral assessments generally take up to 4 hours to complete. This study also uses research EEG. This non-invasive assessment generally takes 30-45 minutes to complete. After the participant's first assessment, he/she will be randomly assigned to receive treatment either immediately or in 6 months, with behavioral assessments throughout. Participants will be involved in the study for a duration of 15-21 months, depending on randomization.

There are no anticipated risks from this study, although it is possible that the participant may react negatively to some of the assessment measures or intervention sessions. For example, at the most extreme, the participant may be fearful of an age-appropriate toy and may cry or physically pull back from the toy. If this should occur, that particular toy presentation, assessment or intervention will be stopped. Sometimes the EEG net can feel uncomfortable, especially if children do not like wearing hats or having anything touch their heads. Because of this, the study team will provide families with the demonstration ("practice") net to use with the participant before his/her session. At any time during the session if the participant becomes too upset or agitated, researchers will stop the session. Loss of confidentiality is a risk of participating in this research study. As described below, researchers will take every measure to keep participation in this research study confidential. Participants may benefit from the intervention by receiving detailed information about your child's cognitive, language, and communication skills both before the intervention begins and after the intervention is completed. Participants also may benefit from the intervention itself, which is aimed at improving social communication skills in infants and toddlers at high risk for neurodevelopmental disorders. Families will receive written feedback on the participants's performance on the behavioral assessments administered during assessment time point 4. These assessments are used for research purposes and therefore are not comprehensive clinical evaluations. Some of the assessments administered will measure social communication skills relevant to Autism Spectrum Disorder (ASD), and the feedback letter will report whether the assessment indicated the possible presence of ASD. The results of the research may also contribute to the broader TSC and autism fields by enhancing the knowledge of the effects of early intervention on social communication skills in TSC. Benefits that participating children may derive from the intervention may lead to greater benefits for all children with autism and/or TSC.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of Tuberous Sclerosis Complex

Exclusion Criteria:

* A mental age less than 6 months. A plan for epilepsy surgery during the study participation period.

Ages: 6 Months to 40 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
ESCS (Early Social Communication Scales) Assessment. | 3 months
  Change from baseline in the amount of time spent in a Joint Attention (the coordination of attention between objects and people for the purpose of sharing) state at 3 months; ESCS is an experimental measure reported as frequency for requesting and joint attention in 15-minute intervals
ESCS (Early Social Communication Scales) Assessment. | 6 months
  Change from baseline in the amount of time spent in a Joint Attention (the coordination of attention between objects and people for the purpose of sharing) state at 6 months; ESCS is an experimental measure reported as frequency for requesting and joint attention in 15-minute intervals
Parent Caregiver Interaction assesses the amount of time the parent and child spend in engaged in the same play routine. | 3 months
  change from baseline in Joint Engagement (shared engagement in a play routine) at 3 months into study participation, according to the parent caregiver interaction assessment.
Parent Caregiver Interaction assesses the amount of time the parent and child spend in engaged in the same play routine. | 6 months
  change from baseline in Joint Engagement (shared engagement in a play routine) at 6 months into study participation, according to the parent caregiver interaction assessment.
Structured Play Assessment (SPA) | 3 months
  Change from baseline in Symbolic Play (types of play and level of play) at 3 months; this is an experimental measure reported as types of behaviors reflecting flexibility and diversity of the child's play level, based on distinct sets of toys that target specific developmental markers of play.
SPA | 6 months
  Change from baseline in Symbolic Play (types of play and level of play) at 6 months; this is an experimental measure reported as types of behaviors reflecting flexibility and diversity of the child's play level, based on distinct sets of toys that target specific developmental markers of play.
Mullen Scales of Early Learning (MSEL) | 3 months
  Measures cognitive ability and language development (baseline to 3 months). The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. The test identifies the subject's strengths and weaknesses and assesses early intellectual development.
Mullen | 6 months
  Measures cognitive ability and language development (baseline to 6 months). The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. The test identifies the subject's strengths and weaknesses and assesses early intellectual development.
Social communication | 3 months
  Change from baseline at 3 months in the amount of Parent use of social communication support strategies Parent use of social communication support strategies as taught by JASPER will be measured by a parent-child interaction assessment.
Social communication | 6 months
  Change from baseline at 3 months in the amount of Parent use of social communication support strategies Parent use of social communication support strategies as taught by JASPER will be measured by a parent-child interaction assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Shafali Jeste, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Boston Children's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Hyde C, Pizzano M, McDonald NM, Nelson CA 3rd, Kasari C, Thiele EA, Jeste SS. A telehealth approach to improving clinical trial access for infants with tuberous sclerosis complex. J Neurodev Disord. 2020 Jan 22;12(1):3. doi: 10.1186/s11689-019-9302-0. PMID 31969108
- See also: Related Info — http://www.JETSstudy.org